CLINICAL TRIAL: NCT05287880
Title: Quantitative Analysis of 18F-FAPI Dynamic PET/CT for Accurate Differential Diagnosis of Metastatic Lymph Nodes of Esophageal Squamous Cell Carcinoma
Brief Title: Quantitative Analysis of 18F-FAPI Dynamic PET/CT for Accurate Differential Diagnosis of MLN of ESCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.FZYX.009
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-06

CONDITIONS: Esophageal Squamous Cell Carcinoma; Benign Lymph Node Neoplasm; Malignant Lymph Node Neoplasm
Keywords: ESCC; BLN; MLN; Dynamic PET/CT; 18F-FAPI
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-N0 stage: Patients with malignant lymph nodes.
  Interventions: Diagnostic Test: Dynamic PET/CT
- N0 stage: Patients without malignant lymph nodes.
  Interventions: Diagnostic Test: Dynamic PET/CT

INTERVENTIONS:
Diagnostic Test: Dynamic PET/CT — After transmission CT scan for subsequent PET data attenuation correction, continual dynamic clinical PET scans were performed in a single bed position immediately after 18F-FAPI intravenously injection (210 ± 30 MBq) in list mode for 60 minutes in supine position, dynamic 48 time frames PET/CT imaging was obtained. And then underwent whole body static PET scan.
  Groups: Non-N0 stage
Diagnostic Test: Dynamic PET/CT — After transmission CT scan for subsequent PET data attenuation correction, continual dynamic clinical PET scans were performed in a single bed position immediately after 18F-FAPI intravenously injection (210 ± 30 MBq) in list mode for 60 minutes in supine position, dynamic 48 time frames PET/CT imaging was obtained. And then underwent whole body static PET scan.
  Groups: N0 stage

SUMMARY:
Patients diagnosed with esophageal squamous cell carcinoma based on clinicopathology, laboratory examination and imaging criteria were selected as the research subjects, and compared with conventional 18F-FDG PET/CT. To evaluate the research value of quantitative analysis of 18F-FAPI PET/CT dynamic imaging in the classification of benign and malignant features of primary esophageal squamous cell carcinoma (ESCC) and lymphatic nodules, lesion localization, outcome and prognosis.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is the eighth most common cancer in the world. Like most other cancers, the occurrence and progression of ESCC is a multi-stage process that closely affects the treatment approach such as endoscopic therapy, surgery, radiotherapy or chemotherapy, and the location of the lesion also affects whether the patient is suitable for surgical resection.Accurate preoperative assessment of lymph node metastasis, disease progression and lesion location is of great significance for early diagnosis and determination of neoadjuvant therapy.

FAP is highly expressed in activated mesenchymal fibroblasts and pericytes in 90% of common human epithelial tumors, as well as in lesions characterized by activation of mesenchymal tissues.The expression of FAP promotes the development of tumors, so inhibiting FAP can slow down the growth of tumors.Currently, several small molecule FAP inhibitors have been functionalized for imaging studies.Studies have shown high uptake of FAPI in sarcoma, esophageal cancer, breast cancer, bile duct cancer, and lung cancer.

Dynamic PET/CT imaging technology with high sensitivity and specificity introduces time parameters while using the fusion technology of PET and CT, providing accurate anatomical positioning in the four-dimensional space and reflecting detailed functional information at molecular level such as functional and metabolic levels.Accurate diagnosis of metastatic lymph nodes of esophageal squamous cell carcinoma can be realized by exploring the kinetic process of various positron probes from entering the body to non-specific distribution and specific distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Esophageal squamous cell carcinoma was diagnosed according to gastroscopy and pathological diagnostic criteria;
2. Age above 18 years old, less than 85 years old, no gender restriction;
3. Untreated patients who have not received surgery, chemotherapy, biotherapy or radiotherapy;
4. Laboratory examination:

(1) General physical condition score ECOG: 0-2; (2) No dysfunction of main organs; (3) Oxygen partial pressure ≥ 10.64kPa; (4) WBC ≥ 4×109 L-1; (5) Routine blood hemoglobin ≥ 9.5 g· DL-1; (6) The absolute count of neutrophils ≥ 1.5×109 L-1; (7) Platelet count ≥ 100×109 L-1; (8) Total bilirubin ≤ 1.5 times the upper limit of normal value; (9) Creatinine ≤ 1.25 times the upper limit of normal value; (10) Creatinine clearance rate ≥ 60 mL ·min-1;

5. Can obtain complete follow-up information, understand the situation of this study and sign the informed consent.

Exclusion Criteria:

1. Has had any other malignant tumor within 5 years;
2. Nursing and/or pregnant women;
3. Patients with severe bleeding tendency;
4. Recent severe hemoptysis, severe cough, dyspnea or patients cannot cooperate;
5. Severe emphysema, pulmonary congestion and cor pulmonale;
6. In the opinion of the Investigator, the subject may not be able to complete the study or comply with the requirements of the study (for administrative or other reasons).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: More than 18 years old and less than 85 years old, no gender limitation, first diagnosis of Esophageal squamous cell carcinoma patients. Patients who must comply with all the inclusion criteria are eligible to participate in this study. However,patients who meet any of the exclusion criteria will not be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of SUVmax between MLN and BLN. | 50 min to 60 min
  Comparison of SUVmax between MLN and BLN.
Comparison of K1 between MLN and BLN. | 0 min to 60 min
  Comparison of K1 of 2TM between MLN and BLN.
Comparison of k2 between MLN and BLN. | 0 min to 60 min
  Comparison of k2 of 2TM between MLN and BLN.
Comparison of k3 between MLN and BLN. | 0 min to 60 min
  Comparison of k3 of 2TM between MLN and BLN.
Comparison of k4 between MLN and BLN. | 0 min to 60 min
  Comparison of k4 of 2TM between MLN and BLN.
Comparison of BP between MLN and BLN. | 30 min to 60 min
  Comparison of BP of LoganREF between MLN and BLN.